CLINICAL TRIAL: NCT03321058
Title: Polymedikations-Check Und Medikamenten-Organisation im Alltag
Brief Title: Polymedication-Check With Insight in Patients' Medication Organisation and Comprehension of Generics
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: University of Basel (Other)
Responsible Party: Principal Investigator, Kurt Hersberger, Prof. Dr., University Hospital, Basel, Switzerland
Other Study IDs: PMC-Medication-Organisation
Record Dates: First submitted 2017-06-01; First posted 2017-10-25 (Actual); Last update posted 2017-10-25 (Actual); Status verified 2017-10

CONDITIONS: Medication Therapy Management; Medication Adherence
Keywords: Drug Substitution; Multicompartment Compliance Aid
MeSH Terms: conditions — Medication Adherence | interventions — Restraint, Physical

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Assessment — Assessment of patients' medication organisation and comprehension of generics

SUMMARY:
Patients using multiple drugs including generics have found different solutions to manage their medication. During a Polymedication-Check (medication review type 2a service in community pharmacies) additional information about the organisation of patients' medication in daily life will be compiled in Swiss community pharmacies. Data will allow to better address patients' needs in their medication organisation and comprehension of generics.

ELIGIBILITY:
Inclusion Criteria:

* at least 4 medicines for at least 3 months
* at least 1 generic drug
* at least 1 medicine of ATC code cardiovascular system (C01-10)

Exclusion Criteria:

* medication provided in Multicompartment Compliance Aid or similar device by specific service (pharmacy, elderly home, home care)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population comprises adults (18 years and older) with at least 4 prescribed medicines which they are taking for at least 3 months. One of those medicines must be a generic drug, one must be prescribed for a cardiovascular condition (ATC C01-10). Patients cannot have their medication provided in a Multicompartment Compliance Aid or a similar device by a specific service like home care, pharmacy or home for elderly.
Sampling Method: Probability Sample
Enrollment: 125 (Actual)
Dates: Start 2017-01-06 (Actual); Primary Completion 2017-10-01 (Actual); Study Completion 2017-10-24 (Actual)

PRIMARY OUTCOMES:
Insight in patients' organisation of polymedication | retrospective 3 months
  Patients organise their multiple medications differently in daily life. The study will investigate the different organisation strategies to get a better understanding of patients' behaviour. The behaviour is assessed with a questionnaire containing 14 questions on the management of medication including single choice, multiple choice and free text questions. As example the number of patients already using a medication organisation system will be assessed, the number of patients using a weekly or daily pillbox will be assessed, and who is filling the medication organisation system.
Insight in patients' comprehension of generics | retrospective 3 months
  Patients have a different comprehension of generics including their advantages and disadvantages. The study will investigate patients' comprehension of generics to get a better understanding of patients' behaviour. The comprehension is assessed with a questionnaire containing 4 questions on the believes about generics including single choice, multiple choice and free text questions. As example the number of patients knowing that they use generics is assessed and the patient's personal opinion on advantages and disadvantages of generics is investigated.

SECONDARY OUTCOMES:
Number of patients using Multicompartment Compliance Aids. | retrospective 3 months
  Assessment of proportion of patients already using Multicompartment Compliance Aids prior to interview.
Number of substitutable medicines. | retrospective 3 months
  Assessment of number of brand name medication which could be substituted by generic medication and willingness of pharmacists to recommend generic medicines.
Swallowing difficulties | retrospective 3 months
  Prevalence of present and/or past swallowing difficulties and coping strategies will be assessed. A specific question (from SWAMECO) on the experienced swallowing difficulties is asked and will be answered on a visual analog scale (0 to 100%). If swallowing-difficulties are present, 2 more questions are asked: Which medication is difficult to swallow and how medication is altered in order to be able to swallow them.
Recommended use of Multicompartment Compliance Aids | retrospective 3 months
  Number of recommended use of Multicompartment Compliance Aids by pharmacists.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Basel, Basel, Canton of Basel-City, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Messerli M, Blozik E, Vriends N, Hersberger KE. Impact of a community pharmacist-led medication review on medicines use in patients on polypharmacy--a prospective randomised controlled trial. BMC Health Serv Res. 2016 Apr 23;16:145. doi: 10.1186/s12913-016-1384-8. PMID 27108410
- [Background] Olsson E, Kalvemark Sporrong S. Pharmacists' experiences and attitudes regarding generic drugs and generic substitution: two sides of the coin. Int J Pharm Pract. 2012 Dec;20(6):377-83. doi: 10.1111/j.2042-7174.2012.00214.x. Epub 2012 Jun 1. PMID 23134096
- [Background] Hakonsen H, Eilertsen M, Borge H, Toverud EL. Generic substitution: additional challenge for adherence in hypertensive patients? Curr Med Res Opin. 2009 Oct;25(10):2515-21. doi: 10.1185/03007990903192223. PMID 19708764
- [Background] Nunney J, Raynor DK, Knapp P, Closs SJ. How do the attitudes and beliefs of older people and healthcare professionals impact on the use of multi-compartment compliance aids?: a qualitative study using grounded theory. Drugs Aging. 2011 May 1;28(5):403-14. doi: 10.2165/11587180-000000000-00000. PMID 21542662